CLINICAL TRIAL: NCT03566290
Title: Phase 2, Open-Label Extension Study to Assess Long-Term Safety and Tolerability of Enobosarm (GTx 024) in Postmenopausal Women With Stress Urinary Incontinence
Brief Title: Study to Assess Long-Term Safety/Tolerability of Enobosarm (GTx 024) in Stress Urinary Incontinence
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Development of investigational product was halted.
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G201004
Record Dates: First submitted 2018-05-30; First posted 2018-06-25 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — ostarine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label Extension, 3 mg GTx-024 (Experimental): Eligible subjects from G201002
  Interventions: Drug: GTx-024

INTERVENTIONS:
Drug: GTx-024 — Study drug is an opaque, white to off-white, size 5, oval Softgel capsule containing the active ingredient GTx-024. Subjects will be required to take one 3 mg Softgel capsule per day.
  Other Names: enobosarm

SUMMARY:
This open-label extension study, for subjects from the G201002 study, will provide additional long-term safety and tolerability data for GTx-024. All subjects in this study will receive GTx-024 3 mg orally, once daily.

ELIGIBILITY:
Inclusion Criteria:

* Be an eligible subject from G201002, where an eligible subject is defined as:

  1. one of the first 225 subjects who were randomly assigned to the placebo group in G201002 and who have completed the required treatment and durability periods of that study, or;
  2. any subject from 226 onwards, who was randomly assigned to any treatment group and who completed the required treatment and follow-up periods of that study
* Be able to read, understand, and provide written, dated, informed consent prior to enrollment in the current study and be likely to comply with the study protocol and communicate with study personnel about AEs and other clinically important information
* Provide written consent to participate in the study within the following timeframes:

  1. for G201002 Subjects 1-225, within 30 days after unblinding of G201002 (subjects who consent to participate in G201003 will be allowed to discontinue from that study and consent to this study upon unblinding of G201002)
  2. for G201002 Subjects 226-493, within 30 days of completing both the treatment and follow-up periods of G201002
* Agree to maintain a stable dose of any medication known to affect lower urinary tract function, including but not limited to anticholinergics, tricyclic antidepressants, beta-3 adrenergic agonists, or α-adrenergic blockers, throughout the duration of the study

Exclusion Criteria:

* Starts any new treatment (medication, pelvic floor physical therapy, or other treatment known to impact the pelvic floor) after completing G201002 that is known or suspected to affect lower urinary tract function, including vaginal rejuvenation
* Subject is currently taking systemic sex-hormone products (excludes intravaginal application of estradiol topical/tablet agents and hormones delivered via vaginal rings)
* Has a current cancer diagnosis (with the exception of nonmelanoma skin cancer) or any history of breast or endometrial cancer
* Has a known history or current episode of:

  1. New York Heart Association Stage ≥ 2 hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg) at screening and/or baseline. Subjects with hypertension that has been treated and controlled with medication for ≥ 2 weeks prior to screening are eligible for participation
  2. Recent myocardial infarction or arterial or venous thromboembolic event (within 1 year) or a history of more than 1 myocardial infarction or arterial or venous thromboembolic event
  3. Cardiac-related syncopal event within the past year
  4. Cardio or cerebral vascular disease requiring surgical intervention (e.g., bypass surgery, angioplasty). For subjects with previous stent placement, please contact the medical monitor
  5. Congestive heart failure of Stage > 2 according to New York Heart Association criteria
  6. Angina pectoris
* Has a current or past history of any physical condition that, in the investigator's opinion, might put the subject at risk, impact the absorption of the study drug, or interfere with interpretation of study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Safety of GTx-024, adverse events | baseline through study completion, an average of 1 year
  Change from baseline in incidence of adverse events
Safety of GTx-024, liver function test | baseline through study completion, an average of 1 year
  Change from baseline in liver function test
Safety of GTx-024, lipid panel | baseline through study completion, an average of 1 year
  Change from baseline in lipid panel
Safety of GTx-024, sex-hormone binding globulin levels | baseline through study completion, an average of 1 year
  Change from baseline in sex-hormone binding globulin levels
Safety of GTx-024, testosterone levels | baseline through study completion, an average of 1 year
  Change from baseline in testosterone levels
Safety of GTx-024, endometrial stripe thickness | baseline through study completion, an average of 1 year
  Change from baseline in endometrial stripe thickness as measured by transvaginal ultrasound
Safety of GTx-024, weight | baseline through study completion, an average of 1 year
  Change from baseline weight

SECONDARY OUTCOMES:
Efficacy of GTx-024, stress incontinence | baseline through study completion, an average of 1 year
  Change from baseline in the mean number of stress incontinence episodes per day
Efficacy of GTx-024, patient global impression of severity | baseline through study completion, an average of 1 year
  Change in patient global impression of severity (PGI-S; scale: 1-normal, 2-mild, 3-moderate, 4-severe; representing severity of urinary tract dysfunction)
Efficacy of GTx-024, patient global impression of improvement | baseline through study completion, an average of 1 year
  Change in patient global impression of improvement (PGI-I; scale: 1-very much better, 2-much better, 3-a little better, 4-no change, 5-a little worse, 6-much worse, 7-very much worse; representing change in urinary tract dysfunction from initiation of therapy)
Efficacy of GTx-024, urge incontinence | baseline through study completion, an average of 1 year
  Change from baseline in the mean number of urge incontinence episodes per day
Efficacy of GTx-024, total incontinence | baseline through study completion, an average of 1 year
  Change from baseline in the mean number of total (stress + urge) incontinence episodes per day

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Professor & Chair, Department of Urology, Oakland University Wm. Beaumont School of Medicine
Locations (46):
- United States (46):
  - Urology Center of Alabama, Homewood, Alabama
  - Coastal Clinical Research Inc, Mobile, Alabama
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Urology Associates Research, Englewood, Colorado
  - Women's Health Specialty Care, Farmington, Connecticut
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - So. Florida Medical Research, Aventura, Florida
  - Tampa Bay Medical Research Inc, Clearwater, Florida
  - Midland Florida Clinical Research Center LLC, DeLand, Florida
  - Medical Research of Florida, Miami, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Mount Vernon Clinical Research LLC, Sandy Springs, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Idaho Urologic Institue, Meridian, Idaho
  - First Urology PSC, Jeffersonville, Indiana
  - Iowa Clinic, West Des Moines, Iowa
  - DelRicht Clinical Research, LLC, New Orleans, Louisiana
  - Regional Urology, Shreveport, Louisiana
  - Chesapeake Urology Associates PA, Hanover, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Bay State clinical Trials, Watertown, Massachusetts
  - Beyer Research, Kalamazoo, Michigan
  - William Beaumont Hospital Urology Research, Royal Oak, Michigan
  - Women's Clinic of Lincoln, Lincoln, Nebraska
  - Sheldon J Freedman MD Ltd, Las Vegas, Nevada
  - Premier Urology Group, LL, Edison, New Jersey
  - Lawrence Obs Gyn clinical Research, Lawrenceville, New Jersey
  - Accumed Research Associates, Garden City, New York
  - Manhattan Medical Research Practice PLLC, New York, New York
  - Premier Medical Group, Poughkeepsie, New York
  - Circuit Clinical, West Seneca, New York
  - American Health Research Inc, Charlotte, North Carolina
  - Eastern Carolina Women's, New Bern, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Aventiv Research, Columbus, Ohio
  - Urologic Consultants of Southeastern PA LLP, Bala-Cynwyd, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - Elligo - Austin Area OBGYN, Austin, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - Urology San Antonio Research PA, San Antonio, Texas
  - Synexus Clinical Research Advantage, Inc. - Wasatch Peak Family Practice, Layton, Utah
  - Urology of Virginia, Virginia Beach, Virginia
  - Seattle Womens: Health, Research, Gynocology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT03566290/Prot_SAP_000.pdf